CLINICAL TRIAL: NCT02138838
Title: A Randomized, Open-label, Controlled Study to Assess the Efficacy and Safety of Cinacalcet HCl in Pediatric Subjects With Secondary Hyperparathyroidism and Chronic Kidney Disease Receiving Dialysis
Brief Title: Efficacy and Safety of Cinacalcet in Pediatric Patients With Secondary Hyperparathyroidism (SHPT) and Chronic Kidney Disease (CKD) on Dialysis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Amgen decided to terminate the study early to be able to meet US regulatory timelines fo filing. Subjects in treatment were rolled over to the 20140159 study.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20130356; 2013-004958-18 (EudraCT Number)
Record Dates: First submitted 2014-04-01; First posted 2014-05-15 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Chronic Kidney Disease, Secondary Hyperparathyroidism
Keywords: Chronic Kidney Disease, Secondary Hyperparathyroidism, Dialysis, Pediatric
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — Cinacalcet; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care therapy included the use of vitamin D sterols, calcium supplementation, and phosphate binders.
  Interventions: Dietary Supplement: Standard of Care
- Cinacalcet (Experimental): In addition to standard of care participants received cinacalcet at a starting dose (based on dry body weight) of 0.20 mg/kg administered once a day by mouth. Dose adjustments and withholding were based on ionized calcium levels, plasma iPTH, and corrected calcium levels.
  Interventions: Drug: Cinacalcet HCl; Dietary Supplement: Standard of Care

INTERVENTIONS:
Drug: Cinacalcet HCl — Capsules were opened and either sprinkled onto soft food (≥ 5 mg dose) or suspended into a sucrose syrup (≥ 2.5 mg dose) to create a liquid suspension for administration. Tablets were used for doses of 30 mg and higher in participants who could swallow tablets.
  Other Names: Sensipar®; Mimpara®
  Arms: Cinacalcet
Dietary Supplement: Standard of Care — Standard of care therapy included the use of vitamin D sterols, calcium supplementation, and phosphate binders.

SUMMARY:
The primary objective was to evaluate the efficacy of cinacalcet for reducing the plasma intact parathyroid hormone (iPTH) level by ≥ 30%.

DETAILED DESCRIPTION:
This was a 24-week, randomized, multicenter, open-label, controlled study. Participants were randomized into one of two treatment arms; oral administration of cinacalcet daily in addition to standard of care treatment, or standard of care alone. Randomization was stratified by age group (6 to < 12 and 12 to < 18 years of age). All participants received standard of care which could include therapy with Vitamin D sterols, calcium supplementation, and phosphate binders.

Participants in both treatment groups who completed the 20-week treatment period and those who ended the study due to study closure were eligible to enroll in an open-label extension study (20140159; NCT02341417) for further safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 - < 18 years
* Diagnosis of SHPT with the mean of the two consecutive central laboratory iPTH values ≥ 300 pg/mL during screening
* Corrected calcium value of ≥ 8.8 mg/dL during screening
* Diagnosis of CKD, receiving either hemodialysis or peritoneal dialysis, for ≥ 30 days prior to screening
* Parent or legally acceptable representative has provided written informed consent and subject has provided written assent when required by institutional guidelines

Exclusion Criteria:

* History of congenital long QT syndrome, second or third degree heart block, ventricular tachyarrhythmias or other conditions associated with prolonged QT interval
* Corrected QT interval (QTc) > 500 ms, using Bazett's formula
* QTc ≥ 450 to ≤ 500 ms, using Bazett's formula, unless written permission to enroll is provided by the investigator after consultation with a pediatric cardiologist
* Use of grapefruit juice, herbal medications, or potent cytochrome P450 3A4 (CYP3A4) inhibitors (eg, erythromycin, clarithromycin, ketoconazole, itraconazole)
* Use of concomitant medications that may prolong the QTc interval (eg, ondansetron, albuterol)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2014-11-07 (Actual); Primary Completion 2016-06-23 (Actual); Study Completion 2016-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (57):
- United States (25):
  - Research Site, Los Angeles, California
  - Research Site, Wilmington, Delaware
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, West Orange, New Jersey
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Research Site, Prague, Czechia
- France (5):
  - Research Site, Bron
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Paris
- Germany (3):
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Marburg
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Szeged
- Italy (3):
  - Research Site, Genova
  - Research Site, Napoli
  - Research Site, Torino
- Research Site, Vilinus, Lithuania
- Research Site, Grafton, Auckland, New Zealand
- Poland (3):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
- Research Site, Porto, Portugal
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Samara
- Research Site, Košice, Slovakia
- Spain (2):
  - Research Site, Barcelona, Catalonia
  - Research Site, Espluques de LLobregat, Catalonia
- Research Site, Kyiv, Ukraine

REFERENCES:
- [Background] Chen P, Sohn W, Narayanan A, Gisleskog PO, Melhem M. Bridging adults and paediatrics with secondary hyperparathyroidism receiving haemodialysis: a pharmacokinetic-pharmacodynamic analysis of cinacalcet. Br J Clin Pharmacol. 2019 Jun;85(6):1312-1325. doi: 10.1111/bcp.13900. Epub 2019 Apr 25. PMID 30756425
- [Background] Warady BA, Ng E, Bloss L, Mo M, Schaefer F, Bacchetta J. Cinacalcet studies in pediatric subjects with secondary hyperparathyroidism receiving dialysis. Pediatr Nephrol. 2020 Sep;35(9):1679-1697. doi: 10.1007/s00467-020-04516-4. Epub 2020 May 4. PMID 32367309
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 32 centers in Belgium, Czech Republic, France, Germany, Greece, Hungary, Lithuania, Poland, Portugal, Russia Federation, Slovakia, Spain, Ukraine, and the United States.
Pre-assignment Details: Eligible participants were randomized to 1 of 2 treatment groups in a 1:1 ratio: cinacalcet daily in addition to standard of care (SOC) therapy or SOC therapy alone. Randomization was stratified by age group (6 to < 12 and 12 to < 18 years). Participants remained on treatment for 20 weeks or until the time of renal transplant or parathyroidectomy.
Period: Overall Study
Arm/Group | Standard of Care | Cinacalcet
Started | 28 | 27
Received Study Drug | 28 | 25
Completed | 20 | 16
Not Completed | 8 | 11
Not completed — Study Closure | 7 | 6
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Cinacalcet | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (3.5) | 12.8 (3.9) | 12.6 (3.6)
Age, Customized [Number; unit: participants]
  6 to < 12 years | 9 | 9 | 18
  12 to < 18 years | 19 | 18 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 13 | 15 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Black (or African American) | 4 | 5 | 9
  White | 23 | 19 | 42
  Mixed Race | 0 | 1 | 1
  Other | 1 | 2 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 4 | 0 | 4
  Not Hispanic/Latino | 24 | 27 | 51
Intact Parathyroid Hormone Level [Mean (Standard Deviation); unit: pg/mL] | 1228.43 (732.08) | 945.72 (635.35) | 1092.31 (695.53)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a ≥ 30% Reduction From Baseline In Mean Plasma iPTH During Weeks 11 to 15
Description: Intact parathyroid hormone (iPTH) levels were measured at weeks 11 and 15; the mean value from these 2 measurements was calculated.
  This endpoint was the primary endpoint in the US only.
Time Frame: Baseline and weeks 11 to 15
Population: The analysis was conducted using the full analysis set; participants who had no week 11 or 15 iPTH values were considered non-responders (non-responder imputation).
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Cinacalcet
Number analyzed (Participants) | 28 | 27
percentage of participants | 17.9 | 25.9
Statistical Analysis 1: Comparison: Standard of Care vs Cinacalcet; Test type: Superiority or Other; p = 0.48, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by baseline age group; Treatment Difference = 8.1, 95% CI 2-sided [-13.7 to 29.9] — SOC+Cinacalcet - SOC

2. Primary Outcome: Percentage of Participants Who Achieved a ≥ 30% Reduction From Baseline in Mean Plasma Intact Parathyroid Hormone During the Efficacy Assessment Period
Description: Intact parathyroid hormone (iPTH) levels were measured at weeks 17, 18, 19 and 20; the mean value from these measurements was calculated.
  This endpoint was specified as the the primary endpoint in all countries except the United States (US). In the US this endpoint was specified as a secondary efficacy endpoint.
Time Frame: Baseline and the efficacy assessment period (EAP), weeks 17 to 20
Population: The full analysis set (all randomized participants) was used for this analysis. For participants with no iPTH values in the EAP, the mean of the last 2 available postbaseline values was used. If only 1 postbaseline value was available, this value was used. If no postbaseline value was available, the participant was considered a non-responder.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Cinacalcet
Number analyzed (Participants) | 28 | 27
percentage of participants | 32.1 | 22.2
Statistical Analysis 1: Comparison: Standard of Care vs Cinacalcet; A hierarchical testing procedure was used to test the primary and biochemical secondary endpoints. The primary endpoint was tested at a 2-sided significance level of 0.05. The secondary endpoints were tested using Holm's method at 0.05 (2-sided) should the primary endpoint achieve a significant result; Test type: Superiority or Other; p = 0.42, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel stratified by baseline age group (6-<12 years, 12-<18 years); Treatment Difference = -9.9, 95% CI 2-sided [-33.3 to 13.4] — SOC+Cinacalcet - SOC

3. Secondary Outcome: Percentage of Participants Who Achieved a Mean iPTH ≤ 300 pg/mL (31.8 Pmol/L) During Weeks 17 to 20
Time Frame: Efficacy assessment period, weeks 17 to 20
Population: This analysis was conducted using the full analysis set. For participants with no iPTH values in the EAP, the mean of the last 2 available postbaseline values was used. If only 1 postbaseline value was available, this value was used. If no postbaseline value was available, the participant was considered a non-responder.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Cinacalcet
Number analyzed (Participants) | 28 | 27
percentage of participants | 17.9 | 7.4
Statistical Analysis 1: Comparison: Standard of Care vs Cinacalcet; Test type: Superiority or Other; p = 0.25, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by baseline age group; Treatment Difference = -10.4, 95% CI 2-sided [-27.7 to 6.8] — SOC+Cinacalcet - SOC

4. Secondary Outcome: Percent Change in iPTH From Baseline to the Mean Value During Weeks 17 to 20
Time Frame: Baseline and weeks 17 to 20
Population: This analysis was conducted using the full analysis set using last value carried forward imputation. Participants with no post-baseline values available were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Standard of Care | Cinacalcet
Number analyzed (Participants) | 27 | 24
percent change | -11.3 (11.10) | 7.7 (11.73)
Statistical Analysis 1: Comparison: Standard of Care vs Cinacalcet; Test type: Superiority or Other; p = 0.23, ANCOVA; Analysis of covariance (ANCOVA) with baseline age group as the covariate; Treatment Difference = 19.0, 95% CI 2-sided [-12.5 to 50.5] — SOC+Cinacalcet - SOC

5. Secondary Outcome: Change in Corrected Serum Calcium From Baseline to the Mean Value During Weeks 17 to 20
Time Frame: Baseline and weeks 17 to 20
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Standard of Care | Cinacalcet
Number analyzed (Participants) | 28 | 24
mg/dL | 0.06 (0.126) | -0.28 (0.135)
Statistical Analysis 1: Comparison: Standard of Care vs Cinacalcet; Test type: Superiority or Other; p = 0.059, ANCOVA; Analysis of covariance (ANCOVA) with baseline age group as the covariate; Treatment Difference = -0.34, 95% CI 2-sided [-0.70 to 0.01]

6. Secondary Outcome: Change in Serum Phosphorus From Baseline to the Mean Value During Weeks 17 to 20
Time Frame: Baseline and weeks 17 to 20
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Standard of Care | Cinacalcet
Number analyzed (Participants) | 26 | 24
mg/dL | -0.09 (0.258) | 0.67 (0.266)
Statistical Analysis 1: Comparison: Standard of Care vs Cinacalcet; Test type: Superiority or Other; p = 0.039, ANCOVA; Analysis of covariance (ANCOVA) with baseline age group as the covariate; Treatment Difference = 0.76, 95% CI 2-sided [0.04 to 1.48] — SOC+Cinacalcet - SOC

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: Two participants who were randomized to the cinacalcet group but did not receive cinacalcet were included in the Standard of Care group for safety analysis.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Standard of Care | Cinacalcet
Serious Adverse Events (participants affected / at risk) | 2/30 | 4/25
Other Adverse Events (participants affected / at risk) | 17/30 | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=30) | Cinacalcet (N=25)
Ileus (Gastrointestinal disorders) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Device dislocation (Product Issues) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renovascular hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=30) | Cinacalcet (N=25)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Precocious puberty (Endocrine disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Lip blister (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 3 | 0
Chills (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Vessel puncture site pain (General disorders) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Gastrointestinal infection (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1
Lip infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood calcium decreased (Investigations) | 1 | 1
Blood parathyroid hormone decreased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Weight increased (Investigations) | 2 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Device occlusion (Product Issues) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Catheter placement (Surgical and medical procedures) | 1 | 1
Catheter removal (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Venous stenosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.